CLINICAL TRIAL: NCT01625377
Title: A National, Multi-center, Randomized, Open Label Study to Evaluate the Efficacy and Safety of Everolimus Combined With Enteric-coated Mycophenolate Sodium Compared to the Standard Treatment Combining Tacrolimus and Enteric-coated Mycophenolate Sodium in de Novo Liver Transplant Recipients
Brief Title: A National Multi-center Randomized, Open Label Study to Evaluate Efficacy and Safety of Everolimus With EC-MPS Compared to Standard Treatment Combination Tacrolimus and EC-MPS in de Novo Liver Transplant Recipients
Acronym: SIMCER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001HFR02; 2012-000137-39 (EudraCT Number)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Liver Transplantation
Keywords: Everolimus,; liver transplantation,; early introduction,; renal function
MeSH Terms: interventions — Tacrolimus; Everolimus; Basiliximab; Mycophenolic Acid; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator): From transplantation to randomization: Basiliximab (40mg) at Day 0 and Day 4 + tacrolimus (C0 6-10 ng/ml) from Day 3-Day 5 + mycophenolic acid 1440 mg/d ± oral corticosteroids. From randomization to month 6 : tacrolimus (C0 6-10 ng/ml) + mycophenolic acid 1440 mg/d ± oral corticosteroids
  Interventions: Drug: tacrolimus; Drug: Basiliximab; Drug: Mycophenolic Acid; Drug: Corticosteroids
- Everolimus (RAD001) (Experimental): From transplantation to randomization: Basiliximab (40mg) at Day 0 and Day 4 + tacrolimus (C0 6-10 ng/ml) from Day 3-Day 5 + mycophenolic acid 1440 mg/d ± oral corticosteroids.
  From randomization to month 6 : everolimus (recommended starting dose of 2 mg/day, then adjusted to achieve the target 6 ≤ C0 ≤ 10 ng/mL, until W24) + mycophenolic acid 1440 mg/d ± oral corticosteroids. The dose of tacrolimus was reduced by 50% twice: at the introduction of everolimus and at week 8 post-transplantation. Tacrolimus had to be finally discontinued in week 12 post-transplantation (by week 16 at the latest).
  Interventions: Drug: tacrolimus; Drug: everolimus; Drug: Basiliximab; Drug: Mycophenolic Acid; Drug: Corticosteroids

INTERVENTIONS:
Drug: tacrolimus — Arm 1 : tacrolimus (C0 6-10 ng/ml) from D3-D5 post-transplantation to month 6 post-transplantation. Arm 2 : tacolimus (C0 6-10 ng/ml) from D3-D5 post-transplantation to 16 weeks post-transplantation at the latest.
  Other Names: Prograf®
Drug: everolimus — Arm 1: no everolimus Arm 2: everolimus (C0 6-10 ng/ml) from randomization to month 6 post-transplantation
  Other Names: Certican® / RAD001
  Arms: Everolimus (RAD001)
Drug: Basiliximab — Basiliximab was supplied to the participating centers as marketed, i.e. in packs containing one vial of 20-mg powder, and water for injection (WFI). 20 mg at D0 and D4
  Other Names: Simulect®
Drug: Mycophenolic Acid — Dose of 1440 mg/day from transplantation to month 6 post- transplantation
  Other Names: Myfortic®
Drug: Corticosteroids — Administration of oral corticosteroid therapy was at the discretion of the centers according to their usual practice

SUMMARY:
The aims of the study was to evaluate the safety and efficacy of early introduction one month post-transplantation of everolimus associated to EC-MPS with tacrolimus discontinuation in de novo liver transplant recipients and to evaluate if it leads to a better renal function 6 month post-transplantation compared to standard treatment associating tacrolimus and EC-MPS.

The renal function was estimated by glomerular filtration rate.

ELIGIBILITY:
Key Inclusion Criteria:

* Man or woman aged 18 years or greater, recipient of a primary liver transplant from a deceased donor with whole or split liver

Key Exclusion Criteria:

* Patient recipient of multiple solid organ or islet cell tissue transplants, or have previously received an organ or tissue transplant
* Recipient of a liver from a living donor or cadaveric non heart beating donor
* ABO incompatible transplant graft
* Transplantation following autoimmune liver hepatitis, primitive sclerosing cholangitis or primitive biliary cirrhosis
* Estimated glomerular filtration rate ≤ 30ml/min at selection
* History of malignancy within the 5 past years, other than non-metastatic basal or squamous cell carcinoma and hepatocellular carcinoma
* Alpha-foeto-protein > 1000 ng/ml (only in case of hepatocellular carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2012-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- France (14):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 188 patients were randomized
Groups:
- Tacrolimus: From transplantation to randomization: Basiliximab (20mg) at Day 0 and Day 4 + tacrolimus (C0 6-10 ng/ml) from Day 3-Day 5 + mycophenolic acid 1440 mg/d ± oral corticosteroids. From randomization to month 6 : tacrolimus (C0 6-10 ng/ml) + mycophenolic acid 1440 mg/d ± oral corticosteroids
- Everolimus (RAD001): From transplantation to randomization: Basiliximab (20mg) at Day 0 and Day 4 + tacrolimus (C0 6-10 ng/ml) from Day 3-Day 5 + mycophenolic acid 1440 mg/d ± oral corticosteroids.
  From randomization to month 6 : everolimus (recommended starting dose of 2 mg/day, then adjusted to achieve the target 6 ≤ C0 ≤ 10 ng/mL, until W24) + mycophenolic acid 1440 mg/d ± oral corticosteroids. The dose of tacrolimus was reduced by 50% twice: at the introduction of everolimus and at week 8 post-transplantation. Tacrolimus had to be finally discontinued in week 12 post-transplantation (by week 16 at the latest).
Period: Overall Study
Arm/Group | Tacrolimus | Everolimus (RAD001)
Started | 95 ("Started" indicates randomized patients.) | 93
Safety Set of Population | 94 | 90
Intent to Treat Population | 93 | 90
Completed | 88 | 71
Not Completed | 7 | 22
Not completed — Death | 1 | 1
Not completed — Administrative Problem | 1 | 1
Not completed — Protocol Violation | 0 | 3
Not completed — Adverse Event | 3 | 16
Not completed — Graft loss | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 1
Not completed — Abnormal laboratory values | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Everolimus (RAD001) | Total
Number analyzed (Participants) | 95 | 93 | 188
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (8.24) | 56.5 (8.59) | 56.0 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 81 | 79 | 160

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Randomization) in Renal Function
Description: Change in renal function was measured by change in glomerular filtration rate (GFR). GFR calculated using the abbreviated modification of diet in renal disease (aMDRD) formula.
  GFR in mL/min/1.73m^2 for men of non-black ethnicity: 186 * [C/88]^-1.154 * [A]^-0.023*G*R ; C = serum creatinine (in μmol/L); A = Age (in years). G = 0.742 when the patient is a women; Otherwise G=1 R= 1.21 when the patient was of black ethnicity; Otherwise R = 1 Baseline was Day 28 visit.
Time Frame: Baseline, Week 24
Population: The Intent to treat (ITT) population included all randomized patients who received at least one dose of study treatment post-randomization and for whom a creatinine value a Day 28 and a posterior value were available. The last observation carried forward (LOCF) is used as imputation of missing data.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
mL/min/1.73m^2 | -13.29 (2.75) | 1.05 (2.81)
Statistical Analysis 1: Comparison: Tacrolimus vs Everolimus (RAD001); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -14.34, 95% CI 2-sided [-21.34 to -7.34]

2. Secondary Outcome: Number of Patients With Treatment Failures
Description: Incidence of treatment failures, assessed with composite criterion including treated biopsy proven acute rejection (tBPAR) with a rejection activity index (RAI) according to Banff classification >3, graft loss or death at 6 months.
  Biopsy proven acute rejection (BPAR) was defined as a clinically suspected acute rejection confirmed by biopsy. The Banff Rejection Activity Index (RAI) comprises 3 components scored from 0 to 3: venous endothelial inflammation; bile duct inflammation damage; and portal inflammation; the scores are combined to an overall score (the RAI) ranging from 0 to 9. An overall score of 0-3 is considered indeterminate, score of 4-5 is mild acute, score of 6-7 is moderate acute , and score of 8-9 is severe acute. Only the episode with the highest total RAI score for each participant was counted.
  The graft was presumed to be lost on the day the patient was registered again on the waiting list, or the day he/she received a new graft.
Time Frame: At week 12 and week 24
Population: The Intent to treat (ITT) population included all randomized patients who received at least one dose of study treatment post-randomization and for whom a creatinine value at Day 28 and a posterior value were available.
Measure: Number; unit: Patients
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
Patients
  week 12, Treatment failures - NO | 91 | 88
  week 12, Treatment failures - YES | 2 | 2
  week 24, Treatment failures - NO | 89 | 81
  week 24, Treatment failures - YES | 4 | 9

3. Secondary Outcome: Number of Patients With Treated or Not Treated Biopsy Proven Acute Rejection (BPAR)
Description: Biopsy proven acute rejection was defined as a clinically suspected acute rejection confirmed by biopsy.
Time Frame: at 12 week and 24 week
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
Patients
  Week 12, Treated BPAR | 2 | 2
  Week 12, Not treated BPAR | 0 | 0
  Week 24, Treated BPAR | 2 | 8
  Week 24, Not Treated BPAR | 0 | 1

4. Secondary Outcome: Number of Patients Reported With Different Categories of Severity of BPAR According to Banff Classification
Description: Biopsy proven acute rejection was defined as a clinically suspected acute rejection confirmed by biopsy.
  The severity of BPAR was categorized as :
  Mild (Banff grade I, RAI = 4 and 5) Moderate (Banff grade II, RAI = 6 and 7) Severe (Banff grade III, RAI = 8 and 9) Banff Rejection Activity Index (RAI) comprises 3 components scored from 0 to 3: venous endothelial inflammation; bile duct inflammation damage; and portal inflammation; the scores are combined to an overall score (the RAI) ranging from 0 to 9. An overall score of 0-3 is considered indeterminate, score of 4-5 is mild acute, score of 6-7 is moderate acute , and score of 8-9 is severe acute. Only the episode with the highest total RAI score for each participant was counted.
Time Frame: at 12 week and 24 week
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
Patients
  Week 12: Mild | 1 | 1
  Week 12: Moderate | 1 | 1
  Week 12: Severe | 0 | 0
  Week 24: Mild | 1 | 5
  Week 24: Moderate | 1 | 3
  Week 24: Sever | 0 | 0

5. Secondary Outcome: Number of Patients With Treated or Untreated BPAR With RAI Score Greater Than 3
Description: Biopsy proven acute rejection (BPAR) was defined as a clinically suspected acute rejection confirmed by biopsy. The Banff Rejection Activity Index (RAI) comprises 3 components scored from 0 to 3: venous endothelial inflammation; bile duct inflammation damage; and portal inflammation; the scores are combined to an overall score (the RAI) ranging from 0 to 9. An overall score of 0-3 is considered indeterminate, score of 4-5 is mild acute, score of 6-7 is moderate acute , and score of 8-9 is severe acute. Only the episode with the highest total RAI score for each participant was counted.
  The patients with treated or untreated BPAR having RAI score > 3 were reported in this end point.
Time Frame: At 24 weeks
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
Patients
  Not Treated BPAR: RAI score >3 | 0 | 0
  Not Treated BPAR: Missing RAI score | 0 | 1
  Treated BPAR: RAI score >3 | 2 | 8

6. Secondary Outcome: Number of Patients With Death or Graft Loss
Description: The graft was presumed to be lost on the day the patient was registered again on the waiting list, or the day he/she received a new graft.
Time Frame: at week 24
Population: as for outcome 2
Measure: Number; unit: Patients
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
Patients
  Graft Loss | 1 | 0
  Death | 1 | 1

7. Secondary Outcome: Change From Baseline (Randomization) in Serum Creatinine
Description: Change in serum creatinine concentrations from baseline (randomization) to week 24 post-randomization was one of the efficacy assessments of renal function.
  Baseline was Day 28 visit.
Time Frame: Baseline, Week 24
Population: The Intent to treat (ITT) population included all randomized patients who received at least one dose of study treatment post-randomization and for whom a creatinine value at D28 and a posterior value were available. The last observation carried forward (LOCF) is used as imputation of missing data.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
µmol/L | 7.2 (36.0) | -1.3 (38.53)

8. Secondary Outcome: Change From Baseline (Randomization) in Urine Protein/Creatinine Ratio
Description: Change in urine protein/creatinine ratio from baseline (randomization) to week 24 post-randomization was one of the efficacy assessments of renal function. Baseline was Day 28 visit.
Time Frame: Baseline, week 24
Population: The Intent to treat (ITT) population included all randomized patients who received at least one dose of study treatment post-randomization and for whom urine protein and creatinine value at day 28 and a posterior value were available. LOCF applied.
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 64 | 61
mg/mmol | -2.3 (27.89) | 21.9 (92.00)

9. Secondary Outcome: Change From Baseline (Randomization) in Creatinine Clearance Estimated Using the Adjusted Cockcroft-Gault Formula
Description: Creatinine clearance by the Cockcroft-Gault formula is computed in mL/min/1.73m^2 from the creatinine clearance in mL/min by multiplying it by 1.73 and dividing it by the body surface area Baseline was Day 28 visit.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
mL/min/1.73m^2 | -9.0 (30.63) | 0.7 (25.65)

10. Secondary Outcome: Change From Baseline (Randomization) in Glomerular Filtration Rate Estimated by Abbreviated Modification of Diet in Renal Disease (MDRD) Formula
Description: Change in glomerular filtration rate was calculated using the MDRD abbreviated formula.
  GFR in mL/min/1.73m^2 for men of non-black ethnicity: 186 * [C/88]^-1.154 * [A]^-0.023*G*R ; C = serum creatinine (in μmol/L); A = Age (in years). G = 0.742 when the patient is a women; Otherwise G=1 R= 1.21 when the patient was of black ethnicity; Otherwise R = 1 Baseline was Day 28 visit.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
mL/min/1.73m^2 | -11.8 (34.01) | 0.1 (32.59)

11. Secondary Outcome: Change From Baseline (Randomization) in Glomerular Filtration Rate Estimated by CKD-EPI Formula
Description: GFR estimated by using the Chronic kidney disease- epidemiology (CKD-EPI) formula:
  eGFR (mL/min/1.73m^2) = 141 * min(C/K,1)^ α * max(C/K,1)^-1.209 * 0.993^A * 1.1018 (if male) * 1.159 (if black) where C = serum creatinine (in mg/dL) ; A = Age (in years); K = 0.7 for women and 0.9 for men; α = -0.329 for women and -0.411 for men. Baseline was Day 28 visit.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 93 | 90
mL/min/1.73m^2 | -6.9 (20.11) | 2.4 (22.18)

12. Secondary Outcome: Number of Patients in Different Stages of Chronic Kidney Diseases According to the K/DOQI Classification System
Description: Kidney disease outcomes quality initiative (K/DOQI) classification is based on glomerular filtration rate (GFR), abbreviated MDRD formula (mL/min/1.73m^2) :
  Stage 1 : GFR >= 90; Stage 2 = GFR was between 60-89; Stage 3 = GFR was between 30-59 ; Stage 4 = GFR was between 15-29; Stage 5 = GFR was < 15 (or dialysis)
Time Frame: At Week 24
Population: ITT population included all randomized patients who received at least one dose of study treatment post-randomization and for whom a creatinine value at D28 and a posterior value were available.
Measure: Number; unit: Patients
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 86 | 74
Patients
  Stage 1 | 24 (27.89) | 41 (92.00)
  Stage 2 | 34 | 29
  Stage 3 | 28 | 4
  Stage 4 | 0 | 0
  Stage 5 | 0 | 0

13. Secondary Outcome: Number of Patients With Any Adverse Events, Serious Adverse Events, Death and Premature Discontinuation
Description: Baseline was Day 28 visit. This endpoint reports patients with total adverse events (any), serious adverse events, death and premature discontinuation.
Time Frame: Baseline to 24 weeks
Population: The safety population included all randomized patients who received at least one dose of study treatment post-randomization and for whom there was a post-treatment safety assessment.
Measure: Number; unit: Patients
Arm/Group | Tacrolimus | Everolimus (RAD001)
Number analyzed (Participants) | 94 | 90
Patients
  Any Adverse events | 85 | 81
  Serious Adverse events | 28 | 42
  Death | 1 | 2
  At least one AE led to premature discontinuation | 4 | 18

ADVERSE EVENTS:
Description: The safety population included all randomized patients who received at least one dose of study treatment post-randomization and for whom there was a post-treatment safety assessment.
Arm/Group | Tacrolimus | Everolimus (RAD001)
Serious Adverse Events (participants affected / at risk) | 28/94 | 42/90
Other Adverse Events (participants affected / at risk) | 68/94 | 64/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=94) | Everolimus (RAD001) (N=90)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Device dislocation (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 2
Generalised oedema (General disorders) | 0 | 1
Hyperthermia (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1
Biloma (Hepatobiliary disorders) | 1 | 0
Cholangiolitis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic artery stenosis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic vein stenosis (Hepatobiliary disorders) | 1 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 0 | 1
Liver transplant rejection (Immune system disorders) | 3 | 5
Transplant rejection (Immune system disorders) | 0 | 2
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 1
Cholangitis suppurative (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Hepatic infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Oral infection (Infections and infestations) | 0 | 1
Pneumococcal infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 5
Septic arthritis staphylococcal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Sinusitis aspergillus (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 4 | 5
Liver graft loss (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 3
Renal failure acute (Renal and urinary disorders) | 2 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Physical disability (Social circumstances) | 0 | 1
Diabetes mellitus management (Surgical and medical procedures) | 1 | 1
Drain removal (Surgical and medical procedures) | 1 | 0
Umbilical hernia repair (Surgical and medical procedures) | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus (N=94) | Everolimus (RAD001) (N=90)
Anaemia (Blood and lymphatic system disorders) | 7 | 12
Leukopenia (Blood and lymphatic system disorders) | 8 | 10
Lymphopenia (Blood and lymphatic system disorders) | 6 | 4
Neutropenia (Blood and lymphatic system disorders) | 14 | 9
Pancytopenia (Blood and lymphatic system disorders) | 1 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 8
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 8
Diarrhoea (Gastrointestinal disorders) | 16 | 6
Oedema peripheral (General disorders) | 6 | 7
Cholestasis (Hepatobiliary disorders) | 12 | 24
Hepatocellular injury (Hepatobiliary disorders) | 4 | 16
Urinary tract infection (Infections and infestations) | 6 | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 11
Renal failure (Renal and urinary disorders) | 11 | 3
Hypertension (Vascular disorders) | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.